CLINICAL TRIAL: NCT04325971
Title: Study of Eye Movements as Markers of the Physiological, Cerebral and Cognitive State of Healthy Subjects
Acronym: EyeProxy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Grenoble Institut des Neurosciences (Other); GIPSA-LAB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC20.063
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — Neuroimaging

STUDY DESIGN:
Masking Description: anonymisation of all data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): All healthy subject are gathered in one arm
  Interventions: Other: Neuroimaging

INTERVENTIONS:
Other: Neuroimaging — MR, EEG recordings

SUMMARY:
The goal of this study is the multimodal exploration via eyetracking, MRI and EEG data of ocular movements and the corresponding brain activation during ecologic visual stimulation in the healthy population.

DETAILED DESCRIPTION:
Cerebral activation following visual stimulation is explored using two neuroimaging techniques EEG and MRI while eye movements are recorded. Three experiments are performed: in MR scanner 1) functional localisation of specific areas: LOC, FFA, MT/V5, V1 and V2 and 2) a saccadic choice experiment; with EEG, replication of the experiments performed in the MR scanner and 3) an additional experiment of movement detection during the ocular saccades.

Thirty young volunteers (18-40 y old) are involved.

ELIGIBILITY:
Inclusion Criteria:

* Normal vision or corrected to normal
* Social security affiliation
* Signed consent to participate
* No pregnancy fo women

Exclusion Criteria:

* Audition and motor troubles
* Incapable to decide (Persons mentioned in L1121-5,6 et 8 of public health code)
* Neurological disorders
* Pathology affecting oculomotor control
* MRI incompatibility

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Eye movement brain networks | 24 months
  Identification of the cerebral locus of ocular movement via MRI & EEG

SECONDARY OUTCOMES:
OculoDB | 24 months
  Database repository of healthy population

CONTACTS AND LOCATIONS:
Overall Officials: Sara MEONI, PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No